CLINICAL TRIAL: NCT06618495
Title: Clinical Study and Molecular Mechanism of Xuesaitong Soft Capsule in the Treatment of Acute Coronary Syndrome After Percutaneous Coronary Intervention
Brief Title: Clinical Study and Molecular Mechanism of Xuesaitong Soft Capsule in the Treatment of Acute Coronary Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024XLA098-2
Record Dates: First submitted 2024-06-28; First posted 2024-10-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; traditional Chinese medicine; Total saponins of Panax notoginseng
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Routine western medicine treatment (oral drug therapy and standard percutaneous coronary intervention) + Xuesaitong soft capsule, 0.33g/ tablets, 2 tablets each time, twice a day. The treatment period is 4 weeks
  Interventions: Drug: Xuesaitong soft capsule (main ingredient is Panax notoginseng saponins)

INTERVENTIONS:
Drug: Xuesaitong soft capsule (main ingredient is Panax notoginseng saponins) — Routine western medicine treatment (oral drug therapy and standard percutaneous coronary intervention) + Xuesaitong soft capsule, 0.33g/ tablets, 2 tablets each time, twice a day. The treatment period is 4 weeks.

SUMMARY:
To evaluate the platelet function, clinical efficacy, prognosis and safety of Xuesaitong soft capsule in the treatment of acute coronary syndrome, 50 patients with acute coronary syndrome after PCI were treated with Xuesaitong soft capsule (mainly Panax notoginseng saponins) for 4 weeks. The macroscopic and microscopic characterization and biological basis of Xuesaitong soft capsule in the treatment of acute coronary syndrome were explained by multi-group techniques (platelet transcription group, metabolic group, protein group).

ELIGIBILITY:
Inclusion Criteria:

* (1) it accords with the diagnostic criteria of western medicine for acute coronary syndrome.

  (2) within 4 weeks after coronary intervention.

  (3) 18 years old ≤ age ≤ 80 years old, male or female.

  (4) voluntarily participate in this clinical trial, give informed consent and sign an informed consent form

Exclusion Criteria:

* (1) uncontrollable hypertension after drug treatment (systolic blood pressure > 180mmHg, or diastolic blood pressure > 110mmHg).

  (2) increased risk of bleeding: previous history of hemorrhagic stroke; intracranial aneurysms; trauma or major surgery within 1 month (including bypass surgery); diseases currently suffering from active bleeding, etc.

  (3) patients with history of digestive tract ulcer and massive gastrointestinal bleeding.

  (4) severe organic heart disease, such as patients with LVEF < 35% or NYHA/Killip cardiac function grade IV.

  (5) those with a history of malignant arrhythmias (arrhythmias affected by hemodynamics, requiring drug or electrical cardioversion, or cardiopulmonary resuscitation), congenital heart disease or malignant tumor were considered unable to participate in the trial.

  (6) severe hepatic and renal insufficiency: glutamic pyruvic transaminase (ALT) or aspartate oxaloacetic transaminase (AST) ≥ 3 × normal upper limit (ULN) or total bilirubin (TBIL) ≥ 2 × ULN; or creatinine clearance (Ccr < 30ml/min).

  (7) Women in pregnancy (defined as positive blood pregnancy test) and lactating women.

  (8) those with a history of blood donation or significant blood loss in the last 3 months (≥ 400ml).

  (9) people with a previous history of alcoholism (i.e. men drink more than 28 standard units per week and women drink more than 21 standard units per week (1 standard unit contains 14g alcohol, such as 360mL beer or 25mL spirits or 150mL wine with 40% alcohol content); or screen those who drink regularly in the first 6 months (that is, more than 14 standard units per week).

  (10) those with a history of drug abuse and drug dependence within one year before screening.

  (11) those who have participated in other clinical trials and taken trial drugs in the past 3 months.

  (12) people who are allergic or intolerant to aspirin or P2Y12 receptor inhibitors.

  (13) those who are allergic to the ingredients of the test drugs.

  (14) other situations in which the researchers think it is not appropriate to participate in this experiment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-11-02 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Transcriptome analysis of patients' platelets collected before and after treatment | 4 weeks
  This measure involves the collection of patients' platelets for comprehensive transcriptome analysis. This analysis aims to identify changes in gene expression profiles before and after treatment. Data will be summarized based on differentially expressed genes, providing insights into the impact of treatment on platelet function at the transcriptional level.
Metabolomics analysis of patients' platelets collected before and after treatment | 4 weeks
  This measure involves the collection of patients' platelets for comprehensive metabolomics analysis. This analysis aims to identify changes in metabolic pathways and metabolites before and after treatment. Data will be summarized based on identified metabolites and altered metabolic pathways, which will help elucidate the treatment's effects on platelet function at the metabolic level.
Proteomics analysis of patients' platelets collected before and after treatment | 4 weeks
  This measure involves the collection of patients' platelets for comprehensive proteomics analysis. This analysis aims to identify changes in protein expression patterns before and after treatment. Data will be summarized based on differentially expressed proteins, providing insights into the treatment's impact on platelet function at the proteomic level.

SECONDARY OUTCOMES:
Changes in platelet granule markers, including platelet factor 4 (PF4) and β-thromboglobulin, before and after treatment, as assessed by ELISA | 4 weeks
  This outcome measure will assess changes in platelet granule markers, including platelet factor 4 (PF4) and β-thromboglobulin, before and after treatment. Both markers will be measured using enzyme-linked immunosorbent assay (ELISA) and reported in consistent units (pg/mL). Data will be summarized based on the change in levels of each marker from baseline to post-treatment, and any significant changes will be noted.
Changes in platelet surface activation markers and platelet-neutrophil aggregation before and after treatment, as assessed by flow cytometry | 4 weeks
  This outcome measure involves the detection of changes in platelet surface activation markers, including P-selectin (CD62P) and the GPIIb/IIIa complex (CD41/CD61), using flow cytometry. Additionally, platelet-neutrophil aggregation will be assessed by measuring the co-expression of CD41 (platelet marker) and CD15 (neutrophil marker). These analyses will quantify the impact of treatment on platelet activation and the interaction between platelets and neutrophils, with results presented as mean fluorescence intensity for each marker. Changes will be compared before and after treatment.
white blood cell count and red blood cell count | 4 weeks
  The white blood cell count and red blood cell count will be measured in cells per microliter (cells/µL). Data will be summarized by the number of participants with values outside the normal reference range, and any significant changes from baseline will be reported.
hemoglobin levels | 4 weeks
  Hemoglobin will be measured in grams per deciliter (g/dL). The number of participants with values outside the normal range will be reported, along with any significant changes from baseline.
hematocrit levels | 4 weeks
  Hematocrit will be reported as a percentage (%), and the number of participants with abnormal values will be summarized.
platelet count | 4 weeks
  Platelet count will be measured in platelets per microliter (platelets/µL). Participants with values outside the normal range will be recorded, along with any significant changes from baseline.
Urine analysis of biochemical markers | 4 weeks
  Urine glucose, protein, and ketones will be measured qualitatively (e.g., negative, trace, 1+, 2+) or quantitatively (e.g., mg/dL). Specific gravity will be measured as a ratio. Data will be summarized by the number of participants with abnormal levels or significant changes from baseline for each parameter.
Urine analysis of cellular components | 4 weeks
  Red blood cells (RBCs), white blood cells (WBCs), and epithelial cells will be measured as the number of cells per high-power field (HPF). Data will be summarized by identifying any abnormal findings (e.g., hematuria or pyuria) or significant changes from baseline.
Stool appearance | 4 weeks
  he consistency and color of stool will be evaluated. Stool color will be categorized (e.g., light brown, green, dark brown), and stool consistency will be assessed on a scale ranging from loose to hard. Data will be presented as categories for stool color and consistency grades.
Biochemical components in stool | 4 weeks
  The presence of blood, mucus, or parasites will be assessed using qualitative measures. Results will be reported as "positive" or "negative" for each component (e.g., blood present: yes/no).
Cellular components in stool | 4 weeks
  Stool will be examined for cellular components such as red and white blood cells. The number of cells per high-power field (HPF) will be recorded and summarized as mean counts (e.g., number of red blood cells/HPF).
liver function based on the enzyme levels | 4 weeks
  Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) will be measured in units per liter (U/L). Data will be summarized by the number of participants with values outside the normal reference range for each enzyme, and significant changes from baseline will be noted.
liver function based on the bilirubin levels | 4 weeks
  Total bilirubin will be measured in milligrams per deciliter (mg/dL). Participants with abnormal bilirubin levels or significant changes from baseline will be reported.
Serum creatinine and blood urea nitrogen (BUN) | 4 weeks
  Both will be measured in milligrams per deciliter (mg/dL). Data will be summarized by the number of participants with levels outside the normal reference range for each parameter, and significant changes from baseline will be noted.
Estimated glomerular filtration rate (GFR) | 4 weeks
  GFR will be estimated and reported in milliliters per minute per 1.73 m² (mL/min/1.73 m²). Participants with abnormal GFR values or significant changes from baseline will be recorded.
Prothrombin time (PT) and activated partial thromboplastin time (aPTT) | 4 weeks
  Both will be measured in seconds (s). Data will be summarized by the number of participants with values outside the normal reference range for each parameter, and significant changes from baseline will be noted.
International normalized ratio (INR) | 4 weeks
  INR will be reported as a unitless value. Participants with abnormal INR values or significant changes from baseline will be recorded.
Assessment of electrocardiogram (ECG) parameters, including QT interval, heart rate, and ST segment changes, before and after treatment | 4 weeks
  This measure involves evaluating various ECG parameters to monitor cardiac electrical activity. Specifically, it includes the measurement of the QT interval, heart rate, and any changes in the ST segment. The ECG recordings will be analyzed before and after treatment to assess the impact on cardiac function. Data will be summarized by the measurement of these parameters and any significant deviations from normal ranges

CONTACTS AND LOCATIONS:
Overall Officials: Dazhuo Shi, professor, Principal Investigator — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Xiyuan Hospital, China Academy of Chinese Medical Sciences, Beijing, China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT06618495/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT06618495/ICF_001.pdf